CLINICAL TRIAL: NCT04024696
Title: An Open-Label, Non-Randomized Clinical Study to Evaluate Pharmacokinetic (PK) Profiles, Safety, and Tolerability of Abexinostat Monotherapy in Patients With Non-Hodgkin's Lymphoma Who Have Failed Standard of Care
Brief Title: A Clinical Study to Evaluate Pharmacokinetics, Safety, and Tolerability of Abexinostat in Chinese Patients
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xynomic Pharmaceuticals, Inc. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XYN-609
Record Dates: First submitted 2019-07-09; First posted 2019-07-18 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — abexinostat

STUDY DESIGN:
Intervention Model Description: Cohort 1: 40 mg BID Cohort 2: 60 mg BID Cohort 3: 80 mg BID
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dosing Cohorts (Experimental): Three (3) dose cohorts are pre-set to include 40 mg BID, 60 mg BID and 80 mg BID,respectively.The pre-set dose group is subject to change during the study and the actual dosage increment is determined by the Data safety Monitoring Committee (DSMC).
  Interventions: Drug: Abexinostat

INTERVENTIONS:
Drug: Abexinostat — Abexinostat Tosylate Tablets

SUMMARY:
This is an open-label, non-randomized clinical study to evaluate the pharmacokinetic (PK) profiles, safety, tolerability and preliminary efficacy of oral abexinostat monotherapy in patients with non-Hodgkin's lymphoma who have failed standard of care, and thereby to determine the pharmacokinetic (PK) parameters, the maximum tolerated dose (MTD), and the recommended phase 2 dose (RP2D) of the oral monotherapy of abexinostat.

DETAILED DESCRIPTION:
This is an open-label, non-randomized clinical study to evaluate the pharmacokinetic (PK) profiles, safety, tolerability and preliminary efficacy of oral abexinostat monotherapy in patients with non-Hodgkin's lymphoma who have failed standard of care, and thereby to determine the pharmacokinetic (PK) parameters, the maximum tolerated dose (MTD), and the recommended phase 2 dose (RP2D) of the oral monotherapy of abexinostat.

Three (3) dose groups are pre-set to include 40 mg BID, 60 mg BID and 80 mg BID,respectively.The pre-set dose group is subject to change during the study and the actual dosage increment is determined by the Data safety Monitoring Committee (DSMC). A total of 12-16 subjects in the RP2D dose group will be required to accept PK blood sampling for the analysis of PK profiles and parameters. The patients will continue treatment until the occurrence of a DLT event, disease progression, intolerant toxicity, withdrawal of ICF, treatment discontinuation determined by the investigator, lost to follow-up, death, or termination of the study, (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis o f non Hodgkin's lymphoma
* Patients with non-Hodgkin's lymphoma who have either failed standard of care or are intolerant/unapplicable to therapy;
* Subject who has no growth factor supportive therapy, transfusion of blood or blood products within 14 days before the enrollment test
* The patient is capable and willing to accept the follow up according to the protocol and signed or provided the ICF signed by the legal representative
* Contraceptive measures , definition of women of childbearing age and contraceptive requirements

Exclusion Criteria:

* Subjects who have received anti tumor therapy and have not recovered from previous toxicity reactions ( toxicity reactions unrecovered to grade 1 as per NCI CTCAE 5.0
* Subjects who received major surgery (excluding diagnostic biopsy)within 28 days prior to the first dose.
* Subjects who received autologous stem cell transplantation within 3 months or allogeneic stem cell transplantation within 6 months prior to the first dose with active graft versus host response at screening
* Subjects with use of prohibited medication within 7 days or less than 5 half lives prior to the first dose (whichever is shorter), see prohibited medication list
* Participated in other interventional clinical trial within 1 month or 5 half life periods prior to the first dose (whichever is longer), except for non intervention clinical trials
* Evidence suggests that there may be human immunodeficiency virus (HIV) infection , or hepatitis C (HCV) hepatitis virus infection PCR RNA positive);
* Uncontrolled systemic infection or infection requiring intravenous injection of antibiotics
* Lymphoma with central nervous system (CNS) involvement
* Subjects with concurrent other malignant tumors in addition to the studied tumor within 2 years prior to the first dosing , except for the controlled skin basal cell carcinoma , cervical carcinoma in situ, ductal carcinoma in situ , and papillary thyroid carcinoma
* Subject is known to be allergic to the components of abexinostat
* Pregnant and lactating subjects
* Upon the investigator's judgment , the subject has any disease or medical condition that is unstable or may affect safety or study compliance , such as uncontrolled hypertension,uncontrolled diabetes, active bleeding , etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Measure AUC at Different Dose Level | Up to 6 month
  Measure Area under the plasma concentration versus time curve (AUC) levels at different dose level
Measure Cmax at Different Dose Level | Up to 6 month
  Measure Peak Plasma Concentration (Cmax at different dose level
Determine the maximum tolerated dose | Up to 6 month
  Determine the maximum tolerated dose based on observed dose-limiting toxicity at different dose levels

SECONDARY OUTCOMES:
Measure Objective Response Rate | Up to 12 Month
  Measure objective response rate in % at the RP2D in patients with non-Hodgkin's lymphoma who have failed standard of care
Measure Duration of Response | Up to 12 Month
  Measure duration of response in months at the RP2D in patients with non-Hodgkin's lymphoma who have failed standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, M.D.; Prof, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (4):
- China (4):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Zhejiang Cancer Hospital, Hangzhou
  - Tianjin Medical University General Hospital, Tianjin
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gui L, Xie Z, Qin Y, Liu P, Yang J, Chen X, Li Z, Tao R, Shi Y. Safety, pharmacokinetics, and efficacy of abexinostat, an novel histone deacetylase inhibitor, in Chinese patients with relapsed/refractory B cell non-Hodgkin lymphoma: a Phase 1 study. BMC Cancer. 2025 May 30;25(1):967. doi: 10.1186/s12885-025-14370-y. PMID 40442628